CLINICAL TRIAL: NCT02912078
Title: Pocket Warming of Epidural Medication to Shorten Onset of Labor Analgesia
Brief Title: Pocket Warming of Epidural Medication
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ling-Qun Hu, Professor-Clinical, Anesthesiology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016H0153
Record Dates: First submitted 2016-05-02; First posted 2016-09-23 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Epidural Anesthesia in Labor and Delivery

STUDY DESIGN:
Intervention Model Description: we propose to conduct a prospective, randomized controlled trial to compare the initiation of labor with room temperature epidural medication (pharmacy-prepared 0.125% Bupivacaine with Fentanyl 2mcg/ml - 10mL) to the same epidural medication that has been pocket warmed for a minimum of 1 hour
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pocket-warmed epidural medication (Experimental): This arm will consist of pocket-warmed epidural medications to be administered per standard protocol to patients randomized to this group; this group is the pocket-warming group.
  Interventions: Other: Pocket-warming
- Room-temperature epidural medication (Active Comparator): This arm will consist of room-temperature epidural medications to be administered per standard protocol to patients randomized to this group. This group has no experimental intervention; standard of care labor epidural.
  Interventions: Other: Standard of Care Labor Epidural

INTERVENTIONS:
Other: Pocket-warming — Pocket-warming of epidural medication
  Arms: Pocket-warmed epidural medication
Other: Standard of Care Labor Epidural — Labor epidural medication administered per standard of care; no pocket warming.
  Arms: Room-temperature epidural medication

SUMMARY:
This study will examine recent claims regarding the beneficial effect of warming epidural medications in order to hasten the onset of labor analgesia.

DETAILED DESCRIPTION:
Studies have shown that warmed epidural medication resulted in a mean analgesic onset of 9.2 minutes as compared to a mean onset of 16 minutes for the same medication at room temperature. Onset time for pain medication during labor is important to a great many participants, thus techniques to shorten analgesic onset are relevant to daily clinical practice. Combined-spinal epidural (CSE) techniques have been used to improve the onset and reliability of labor analgesia compared to epidural techniques; however, CSEs have risks associated with their usage. Firstly, is not always possible to administer a spinal dose despite successful loss-of resistance with CSE techniques, providing less satisfactory labor analgesia, and secondly, the CSE technique has been associated with a greater incidence of non-reassuring fetal heart tones (FHT), uterine hyperactivity, maternal pruritis, and greater incidence of neurologic sequelae compared to epidural analgesia. Further, CSE labor analgesia is more likely to result in prolonged FHT decelerations if there is FHT abnormalities prior to the neuraxial procedure. Given these potential limitations of CSE techniques for labor analgesia, epidural medication warming may represent an effective alternative for safe and satisfactory labor analgesia.

Previous studies in obstetric and non-obstetric patients undergoing surgery have demonstrated a more rapid onset of sensory blockade in patients receiving body temperature (37 °C) epidural medication compared to room temperature medication, though other reports have found no significant difference in the onset of sensory blockade when comparing body temperature to room temperature epidural medications. To the knowledge of the investigators, there are few studies examining the effect of warmed epidural medications for patients receiving epidural labor analgesia.

In the experience of the investigators' colleagues, the close proximity to the body has a warming effect on the epidural medication and ultimately leads to quicker onset of pain relief once administered. Pocket warming does not warm the medications to the same extent as an incubator, but is certainly less expensive and is readily available to every obstetric anesthesia practice.

The investigators have previously measured the temperature of five 10mL syringes of normal saline at room temperature and at baseline the average was 21.7 °C (range 21.5-21.9 °C), and increased to an average of 29.7 °C (range 29.1 - 30.2 °C) after 1.5 hours of pocket warming. It has not been studied and is unknown if this degree of warming would be effective in enhancing the onset of labor analgesia, but such information is valuable given that an approximate 30 °C temperature may be accomplished by simple pocket warming and is within manufacturer recommended storage temperatures of 15-30 °C.

The investigators also assessed the potential for epidural medication cooling by measuring the temperature of one of the investigator's 10mL saline syringes for twenty minutes after removal from the warm pocket environment. The initial temperature of 30.0 °C had cooled to 27.0 °C by five minutes, 24.7 °C by ten minutes, 22.9 °C by fifteen minutes, and had returned to baseline room temperature by twenty minutes. The time between medication removal and dosing is important to consider given that significant cooling may occur and negate any potential benefits of warming the medication. This cooling effect makes use of a centralized warmer less promising, as it could take 10-20 minutes to position the patient and complete placement of the epidural catheter prior to dosing the medication. The use of a bedside incubator or a pocket warming technique would be useful in this regard, because the medication could be administered immediately after removal from the warm environment.

The investigators hypothesize that pocket warming in the front, upper pocket would be beneficial in enhancing onset of labor analgesia relative to room temperature medication.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a single vertex presentation fetus at term (38-42 weeks)
2. Intact fetal membranes or membrane rupture <6 hours previously
3. Request to have an epidural for labor analgesia
4. Provide written consent for the study.

Exclusion Criteria:

1. Patients being treated/managed for chronic pain
2. Allergies or significant adverse reactions to local anesthetic or opioid medications
3. Contraindication to labor epidural placement
4. Patients with history of spine abnormalities or spine surgery
5. Clinical signs or symptoms of infection
6. Baseline temperature > 37.6 °C
7. Non-English speaking
8. Prisoners
9. Age less than 18 years old

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time until pain score less than or equal to 3 | duration of labor and delivery
  Assess pain level regularly during labor

SECONDARY OUTCOMES:
Labor analgesia satisfaction | first hour of epidural administration
  Patients will assess initiation of labor analgesia using a 1-100 point rating scale at their routine follow-up visit.
Vital Signs | during labor and delivery
  oral temperature, fever (temperature greater than 38 °C), nausea, vomiting, shivering, and blood pressure will be measured during the first 60 minutes of labor analgesia. Fever at any time during labor will be recorded.
Breakthrough pain | during labor
  number of required rescue epidural boluses, time until first manual epidural rescue bolus, and total number of manual anesthetic interventions to treat inadequate labor analgesia will be recorded during labor
Mode of delivery | Delivery
  Mode of delivery will be recorded (i.e. cesarean, spontaneous vaginal or instrumental vaginal delivery)

CONTACTS AND LOCATIONS:
Overall Officials: John Coffman, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No